CLINICAL TRIAL: NCT04364529
Title: Impact of Pit Crew Resuscitation Model on Advanced Life Support Skills in a Simulated Setting: a Randomized Controlled Trial
Brief Title: Implementation of Pit Crew Resuscitation Model on the Training of Advanced Life Support: a Randomized Controlled Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Collaborators: Turku University of Applied Sciences (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: T212/2016
Record Dates: First submitted 2020-03-04; First posted 2020-04-28 (Actual); Last update posted 2021-11-12 (Actual); Status verified 2021-11

CONDITIONS: Advanced Cardiac Life Support
Keywords: non-technical skills; technical skills; Simulation Training; Patient simulation; CRM; Crew Recourse Management; team work; human factors; pit crew model

STUDY DESIGN:
Intervention Model Description: The students are divided into 26 four-person resuscitation teams: one medical student, one student paramedic and two student nurses. These 26 teams are randomidez in two study arms: intervention (pit-crew group) and the control Group.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The partisipants are unknown of the study design. They are told that they have been randomized in two groups who receive ALS education in two different ways.
  Two senior anesthetists analyse the ALS-performance of the video recordings. They are unaware of the study design. They analyze the videos independently and in random order.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (pit crew model group) (Experimental): 13 groups being taught the pit crew model
  Interventions: Other: The pit crew model
- control (traditional ALS education) (No Intervention): 13 groups being taught along traditional ALS education

INTERVENTIONS:
Other: The pit crew model — The pit crew model
  Arms: Intervention (pit crew model group)

SUMMARY:
In this study, a pit crew model is implemented in advanced life support (ALS) simulation training to student groups. The hypothesis is that the tactic model could help to maintain the CPR skills during the six month follow-up period.

DETAILED DESCRIPTION:
Introduction

Technical skills (TS) and non-technical skills (NTS) are two sets of skills required by Crisis resource management (CRM). Sudden cardiac arrest is a time-critical emergency situation in which both skills are needed - it's handled by a team rather than by individual health-care workers.

Because of the relatively rare nature of cardiac arrests in many wards and clinics, regular resuscitation training is necessary. However, the main part of the training is traditionally emphasized to technical skills. The recent research findings of the authors suggest that the TS and NTS seem to associate in a real life resuscitation. The authors wanted to investigate if pre-allocated tasks and positions (a pit crew model) helps to perform better ALS performance and helps to maintain the skills in simulated ALS situations.

Simulation-based education (SBE) is a key tool for teaching CPR. It has demonstrated its effectiveness in promoting skill acquisition and has been suggested as an ideal tool for teaching medical skills allowing learners to engage actively in their learning process while doing no harm to their patients but its effectiveness on improving anesthesiologists NTS is unclear as the matter has not been studied. SBE is particularly good method to create trainees a realistic medical crisis situation (scenario) created within a physical space (simulator) replicating the real environment where trainees goal is to solve the problem, do the diagnose and treat the patient. Afterwards, the simulation debriefing is an crucial part of the whole letting trainees and the instructor to finish the learning process. Traditionally such training has been a standard in professions characterized by high risk caused by 'human factor' such as in aviation and other high risk industries. On the other hand the benefit for maintaining resuscitation skills learned after single SBE is modest thus short - only a few minutes a week - but frequent SBE appears to facilitate transfer of new knowledge and skills into clinical practice. SBE has been shown to improve the satisfaction of learners and skill performance in the simulated environment but it's still unclear whether it improves the patient outcome. Simulation training is expensive though so other teaching methods like mental practice and e-learning could be useful alongside it.

Catchpole and colleagues aimed to improve the quality and safety of handover of pediatric patients from surgery to intensive care using the analogy of a Formula 1 pit stop and expertise from aviation. They introduced a new handover protocol which led to improvements in all aspects of the critical situation. Based on he same idea, a novel resuscitation tactic model (a pit crew model) was developed which predetermines the roles and responsibilities of each resuscitation team members.

Purpose and hypothesis

In this study, advanced life support (ALS) skills are trained to medical students (26 persons), student nurses (52 persons) and student paramedics (26 persons). A pit crew model is taught for every other four-person resuscitation team (intervention group) and for every other group not (control group). The hypothesis is that the pit crew model could improve the quality of advanced life support immidiately after the ALS education (primary outcome) and help to maintain the ALS metrics during the follow-up period (secondary outcome). Additionally, we analyze if the pit-crew model help team physician to take hands free earlier.

Methods

The students are divided into 26 four-person resuscitation teams: one medical student, one student paramedic and two student nurses. Each resuscitation team participates on an ALS course which is based on the 2015 European (the test group) Guidelines for Resuscitation. The participants are randomized in two study arms: intervention and control. The intervention group receives ALS education according the pit crew model while the control Group received traditional ALS training. In the end of the ALS course, the resuscitation team performs a simulated resuscitation situation which is video-recorded. The TS and NTS are later analyzed by the medical professionals using detailed instrument. The hands-on ratio and the time when the team physician takes hands-free analyzed visually from the videos. Later, after six months of the ALS course, the participants will run through a simulated CPR-situation again and the data will be collected as the the same way.

The primary outcome was the difference in the total assessment score between the intervention and control groups after 6-months follow-up. The secondary outcome was the difference in ALS skills after 6-months follow-up.

Ethics The study protocol was approved by the Ethics Committee of Turku University (31/2016).

ELIGIBILITY:
Inclusion Criteria:

* medical student (fourth or fifth year)
* paramedic student (third or fourth year)
* nurse student (third or fourth year)
* participated simulated ALS-situations e.g. in school before

Exclusion Criteria:

* participated more than two real-life ALS-situations

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2017-08-14 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
The difference in the total assessment score between the intervention and control groups after 6-months follow-up. | 6 months follow-up
  The NTS and TS are evaluated with a valid measurement tool developed for this purpose by two independent evaluators. The instrument consist of 59 items (28 items for TS and the rest for NTS) and the scale of +2 to -2 is used. Additionally, raters gave a total assessment score of performance on a scale from 0 to 10 (0=poor, 10=excellent)

SECONDARY OUTCOMES:
The difference in ALS skills after 6-months follow-up. | 6 months follow-up
  The NTS and TS are evaluated with a valid measurement tool developed for this purpose by two independent evaluators. The instrument consist of 59 items (28 items for TS and the rest for NTS) and the scale of +2 to -2 is used.

OTHER OUTCOMES:
Team physician hands-free from the hands-on work and the chest compression hands-on ratio (hands-on time divided by the total ALS time) between the groups. | Baseline and 6 months
  These are calculated visually from the videos.

CONTACTS AND LOCATIONS:
Locations (1):
- Turku University, Turku, Finland

IPD SHARING:
Plan to Share IPD: No
Participants in the videos can be recognized. Video material can not be shared due to patient privacy. Other data is possible to share.

REFERENCES:
- [Background] Cheng A, Auerbach M, Hunt EA, Chang TP, Pusic M, Nadkarni V, Kessler D. Designing and conducting simulation-based research. Pediatrics. 2014 Jun;133(6):1091-101. doi: 10.1542/peds.2013-3267. Epub 2014 May 12. PMID 24819576
- [Background] Rovamo L, Nurmi E, Mattila MM, Suominen P, Silvennoinen M. Effect of a simulation-based workshop on multidisplinary teamwork of newborn emergencies: an intervention study. BMC Res Notes. 2015 Nov 12;8:671. doi: 10.1186/s13104-015-1654-2. PMID 26563963
- [Background] Cheng A, Lang TR, Starr SR, Pusic M, Cook DA. Technology-enhanced simulation and pediatric education: a meta-analysis. Pediatrics. 2014 May;133(5):e1313-23. doi: 10.1542/peds.2013-2139. Epub 2014 Apr 14. PMID 24733867
- [Background] Eppich WJ, Nypaver MM, Mahajan P, Denmark KT, Kennedy C, Joseph MM, Kim I. The role of high-fidelity simulation in training pediatric emergency medicine fellows in the United States and Canada. Pediatr Emerg Care. 2013 Jan;29(1):1-7. doi: 10.1097/PEC.0b013e31827b20d0. PMID 23283253
- [Background] Asarbakhsh M, Sandars J. E-learning: the essential usability perspective. Clin Teach. 2013 Feb;10(1):47-50. doi: 10.1111/j.1743-498X.2012.00627.x. PMID 23294744
- [Background] Didwania A, McGaghie WC, Cohen ER, Butter J, Barsuk JH, Wade LD, Chester R, Wayne DB. Progress toward improving the quality of cardiac arrest medical team responses at an academic teaching hospital. J Grad Med Educ. 2011 Jun;3(2):211-6. doi: 10.4300/JGME-D-10-00144.1. PMID 22655144
- [Background] Wayne DB, Didwania A, Feinglass J, Fudala MJ, Barsuk JH, McGaghie WC. Simulation-based education improves quality of care during cardiac arrest team responses at an academic teaching hospital: a case-control study. Chest. 2008 Jan;133(1):56-61. doi: 10.1378/chest.07-0131. Epub 2007 Jun 15. PMID 17573509
- [Background] Lorello GR, Hicks CM, Ahmed SA, Unger Z, Chandra D, Hayter MA. Mental practice: a simple tool to enhance team-based trauma resuscitation. CJEM. 2016 Mar;18(2):136-42. doi: 10.1017/cem.2015.4. Epub 2015 Apr 10. PMID 25860822
- [Background] Nicastro E, Lo Vecchio A, Liguoro I, Chmielewska A, De Bruyn C, Dolinsek J, Doroshina E, Fessatou S, Pop TL, Prell C, Tabbers MM, Tavares M, Urenden-Elicin P, Bruzzese D, Zakharova I, Sandhu B, Guarino A. The Impact of E-Learning on Adherence to Guidelines for Acute Gastroenteritis: A Single-Arm Intervention Study. PLoS One. 2015 Jul 6;10(7):e0132213. doi: 10.1371/journal.pone.0132213. eCollection 2015. PMID 26148301
- [Background] Catchpole K, Mishra A, Handa A, McCulloch P. Teamwork and error in the operating room: analysis of skills and roles. Ann Surg. 2008 Apr;247(4):699-706. doi: 10.1097/SLA.0b013e3181642ec8. PMID 18362635
- [Background] Mduma E, Ersdal H, Svensen E, Kidanto H, Auestad B, Perlman J. Frequent brief on-site simulation training and reduction in 24-h neonatal mortality--an educational intervention study. Resuscitation. 2015 Aug;93:1-7. doi: 10.1016/j.resuscitation.2015.04.019. Epub 2015 May 6. PMID 25957942
- [Background] Gjeraa K, Moller TP, Ostergaard D. Efficacy of simulation-based trauma team training of non-technical skills. A systematic review. Acta Anaesthesiol Scand. 2014 Aug;58(7):775-87. doi: 10.1111/aas.12336. Epub 2014 May 14. PMID 24828210
- [Background] Issenberg SB, McGaghie WC, Petrusa ER, Lee Gordon D, Scalese RJ. Features and uses of high-fidelity medical simulations that lead to effective learning: a BEME systematic review. Med Teach. 2005 Jan;27(1):10-28. doi: 10.1080/01421590500046924. PMID 16147767